CLINICAL TRIAL: NCT06325891
Title: Microbiota Diversity and Composition in Gastric Cancer by Gastric Mucosal Brushing: a Cross-sectional Case-control Study
Brief Title: Microbiota in Gastric Cancer by Gastric Mucosal Brushing
Status: Recruiting | Type: Observational
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Associate Professor, King Chulalongkorn Memorial Hospital
Other Study IDs: RP025
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
Keywords: Microbiota; Gastric cancer; Mucosal brushing; Mucosal biopsy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Gastric mucosa by gastric mucosal brushing and gastric mucosal biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric cancer group: * Adult patients (≥18 years of age) and undergoing esophagogastroduodenoscopy
  * Patients with pathological diagnosis of high-grade dysplasia or gastric cancer
  Interventions: Diagnostic Test: Gastric mucosal brushing; Diagnostic Test: Gastric mucosal biopsy
- Control group: * Adult patients (≥18 years of age) and undergoing esophagogastroduodenoscopy
  * Patients with no or minimal upper GI symptoms and current EGD appear normal or minimal gastritis
  Interventions: Diagnostic Test: Gastric mucosal brushing; Diagnostic Test: Gastric mucosal biopsy

INTERVENTIONS:
Diagnostic Test: Gastric mucosal brushing — Gastric mucosal brushing will be performed at body of stomach in control group and non-tumorous area of body in gastric cancer group. If gastric body area could not feasible (eg. tumor involvement), then gastric antrum and more proximal part of body will be sampling.
Diagnostic Test: Gastric mucosal biopsy — Gastric mucosal biopsy will be performed at the area within 2 cm. from brushing site.

SUMMARY:
Many studies have shown a significant change of diversity and composition in gut microbiota across the gastric carcinogenesis process, particularly in patients with gastric cancer. However, there has been no analysis of gastric microbiota using the mucosal brushing technique, despite its favoring benefit in microbiota study. Therefore, this study aims to evaluate microbiota profile in patients with gastric cancer, compared to those without gastric cancer by using mucosal brush sampling. This will improve current knowledge of the potential role of the microbiome in patient gastric cancer as a future biomarker marker using brushing sampling.

DETAILED DESCRIPTION:
* Gut microbiota play role in mucosal immune response and strength gut integrity. The dysbiosis or imbalance of microbiota changes microecology and activates the inflammation in gastrointestinal mucosa. It also has been implicated in gastric carcinogenesis.
* Up to date, many studies have shown a significant change of diversity and composition in gut microbiota across the gastric carcinogenesis process, particularly in patients with gastric cancer. Although, Helicobacter pylori infection is potential class I carcinogen in initial step of gastric carcinogenesis, only between 1% and 3% of patient with H. pylori infection develop gastric cancer. In addition, many current studies have revealed significant change in microbiome profile of patient with H. pylori-negative gastric cancers. Many studies have revealed significant change in microbiome profile of patient with H. pylori-negative gastric cancers. Therefore, the investigators have hypothesized that unidentified non-H. pylori bacteria play a role in gastric cancer development.
* However, most of current studies of gastric microbiota in patients with gastric cancer have been conducted in Eastern Asia, particularly in China and Korea, there is still no published data from Thailand. Moreover, all previous studies have used gastric tissue biopsy method. There has been no analysis of gastric microbiota using the mucosal brushing technique, despite its favoring benefit in microbiota study
* This study is pilot phase, cross-sectional and case-control study that aims to evaluate microbiota profile in patients with gastric cancer, compared to those without gastric cancer by using mucosal brush sampling.
* According to previous studies, H. pylori had significant impact on the composition of gastric microbiota. Presence of H. pylori could affect the result of the study. Therefore pre-specified subgroup analysis of H.pylori infection and non-H.pylori infection will be perform.
* Study protocol include
* Age, gender, BMI, smoking history, history of PPI use within 3 months, history of infection within 2 weeks, history of antibiotic use within 3months, history of probiotic use within 3months, history of intraabdominal surgery, history of dietary supplement and herbal use will be recorded in case record form.
* After consent, standard EGD will be performed.
* The gastric mucosa using mucosal brushing with sterile sheathed brush, gastric mucosal biopsy by standard forceps biopsy and rapid urease test for evaluate H.pylori status will be done respectively.
* The gastric mucosal specimen will be keep in sterile tube and immediate keep in freezing at -80C (allow room temperature <2 hr) for 16sRNA sequencing analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age) and undergoing esophagogastroduodenoscopy (EGD)
* Gastric cancer group: patients with pathological diagnosis of high-grade dysplasia or gastric cancer
* Control group: patients with no or minimal upper GI symptoms and current EGD appear normal or minimal gastritis
* Informed consent obtained

Exclusion Criteria:

* Had a history of GI or hepatobiliary surgery
* Had a history of recent (within 4 weeks) antibiotic or probiotic use
* Had a history of PPI use within 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Gastric cancer group: patients with pathological diagnosis of high-grade dysplasia or gastric cancer
  * Control group: patients with no or minimal upper GI symptoms and current EGD appear normal or minimal gastritis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome analysis using gastric mucosal brushing | Through study completion, estimated 1.5 yr
  Gastric mucosal-associated microbiota in patients with gastric cancer and those without gastric cancer using mucosal brush sampling by 16S rRNA sequencing. Including microbiota diversity and composition.

SECONDARY OUTCOMES:
Microbiome analysis using gastric mucosal biopsy | Through study completion, estimate 1.5 years
  Gastric mucosal-associated microbiota between samples obtained from gastric mucosal tissue biopsy and mucosal brushing in patients with gastric cancer and those without gastric cancer

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - King Chulalongkorn memorial hospital, Bangkok